CLINICAL TRIAL: NCT01404429
Title: Randomized Controlled Trial of Two Different Starting Doses of Methotrexate in Rheumatoid Arthritis
Brief Title: Study of Two Different Starting Doses of Methotrexate When Starting Treatment in Rheumatoid Arthritis
Acronym: DMIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Varun Dhir, Assistant Professor, Internal Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKG/992
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Active
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate 7.5 mg per week (Active Comparator)
  Interventions: Drug: Methotrexate
- Methotrexate 15 mg per week (Experimental)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Different doses for both arms followed by similar escalation (2.5 mg every 15 d) till max of 25 mg per week or 3 months completed
  Other Names: MEXATE

SUMMARY:
To use different starting doses of methotrexate (7.5 mg per week) versus 15 mg per week in patients with rheumatoid arthritis, followed by similar hiking up of dose (2.5 mg per 2 weeks, till max of 25 mg per week). To look at the effect on efficacy ( or speed of efficacy) versus the adverse effects.

Hypothesis: There will be no difference in the adverse effects, but better and faster control of disease when starting with a higher methotrexate dose

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis fulfilling the ACR 1987 criteria
* Between 18 years to 65 year of age
* Having active disease Disease activity score (28 joints) DAS28-3 more than 5.1
* Not on methotrexate in the last 2 months
* Permitted to be on corticosteroids if the dosages stable for at least 1 weeks before randomization and if corticosteroid dosage less than 10 mg/day
* Permitted to be on other disease modifying anti-rheumatic drug (DMARD) like sulfasalazine, leflunomide and hydroxychloroquine, if dosages stable for at least 2 weeks before randomization

Exclusion Criteria:

* Pregnant/Breastfeeding
* Ongoing/Recent treatment with methotrexate (2 months)
* Chronic liver disease
* Renal failure
* Any leucopenia or thrombocytopenia
* Breast-feeding
* Desirous of pregnancy in the next 6 months
* Known Hepatitis B or C positive
* Known clinically relevant chronic lung disease: ILD
* Tuberculosis or other active infections
* Known HIV positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New OPD Block, Rheumatology Clinic, Level 3, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Dhir V, Singla M, Gupta N, Goyal P, Sagar V, Sharma A, Khanna S, Singh S. Randomized controlled trial comparing 2 different starting doses of methotrexate in rheumatoid arthritis. Clin Ther. 2014 Jul 1;36(7):1005-15. doi: 10.1016/j.clinthera.2014.05.063. Epub 2014 Jun 26. PMID 24976447
- See also: published manuscript — http://dx.doi.org/10.1016/j.clinthera.2014.05.063

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate 7.5 mg Per Week: Patients started on 7.5 mg of oral methotrexate (weekly) increased by 2.5 mg every 2 weeks (max 25mg weekly)
- Methotrexate 15 mg Per Week: Patients started on 15 mg of oral methotrexate (weekly) increased by 2.5 mg every 2 weeks (max 25mg weekly)
Period: Overall Study
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Started | 47 | 53
Completed | 38 | 46
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Methotrexate 7.5 mg Per Week: Patients started on 7.5 mg of oral methotrexate (weekly) which was then escalated by 2.5 mg every 2 weeks (max 25 mg weekly)
- Methotrexate 15 mg Per Week: Patients started on 15 mg of oral methotrexate (weekly) which was then escalated by 2.5 mg every 2 weeks (max 25 mg weekly)
- Total: Total of all reporting groups
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.3) | 42.8 (11.2) | 43.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the DAS28-3 (Disease Activity Score Using 28 Joints and Using 3 Variables) - Difference Between This Score at 12 Weeks and This Score at Baseline
Description: DAS28-3 is disease activity score using 28 joints and using 3 variables (tender and swollen joint count for 28 joints and ESR(westergren 1st hour) It ranges from 0 to 9.3 where a lower value implies lower disease activity
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Number analyzed (Participants) | 47 | 53
units on a scale | -0.47 (0.86) | -0.55 (0.79)
Statistical Analysis 1: Comparison: Methotrexate 7.5 mg Per Week vs Methotrexate 15 mg Per Week; Test type: Superiority or Other; p = 0.6, t-test, 2 sided; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.26 to 0.54]

2. Primary Outcome: Patients With Good Response (Final DAS28-3 Less Than 3.2 and Fall More Than 1.2)
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Number analyzed (Participants) | 47 | 53
participants | 0 | 1

3. Secondary Outcome: Proportion of Patients Who Withdrew Because of Any Cause
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Number analyzed (Participants) | 47 | 53
participants | 9 | 7

4. Secondary Outcome: Proportion Requiring Stoppage/Decrease/Inability to Hike MTX Due to Cytopenia or Transaminitis (SGOT or SGPT More Than 80IU)
Time Frame: 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Proportion Who Withdrew Due to Intolerance
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Number analyzed (Participants) | 47 | 53
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Methotrexate 7.5 mg Per Week | Methotrexate 15 mg Per Week
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/53
Other Adverse Events (participants affected / at risk) | 9/47 | 22/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate 7.5 mg Per Week (N=47) | Methotrexate 15 mg Per Week (N=53)
Nausea and vomiting (Gastrointestinal disorders) | 9 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No